CLINICAL TRIAL: NCT05675618
Title: Golfing After Orthopaedic Surgery: a Longitudinal Follow-up (GOLF) Project
Brief Title: Return to Golf After Orthopaedic Surgery
Status: Recruiting | Type: Observational
Sponsor: Hospital for Special Surgery, New York (Other)
Collaborators: Royal Infirmary of Edinburgh (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-0437
Record Dates: First submitted 2022-12-28; First posted 2023-01-09 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Hip Osteoarthritis; Knee Osteoarthritis; Shoulder Osteoarthritis
Keywords: return to golf, arthroplasty
MeSH Terms: conditions — Osteoarthritis, Hip; Osteoarthritis, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The GOLF study is a multicenter, prospective study with the goal to investigate golfers' return to the sport following hip, knee or shoulder arthroplasty. The prevalence of return to golf, by level of returning to golf will be assessed at 6 weeks, 3 months, 6 months, and 12 months postoperatively. Patients who are active golfers undergoing joint replacement will be identified from outpatient clinics and pre-assessment clinics and given information about the study at least two weeks prior to surgery. Participants in this study must have a desire to return to golf after surgery. Previous studies have only been able to report the return to golf after arthroplasty retrospectively; the prospective nature of this study will allow for a greater understanding of this process.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+ years
* A self-reported golfer
* Able to consent to treatment
* Indicated for one of the following surgical procedures: total hip arthroplasty, hip resurfacing, revision hip arthroplasty, total knee arthroplasty, unicompartmental knee arthroplasty, revision knee arthroplasty, total shoulder arthroplasty, reverse shoulder arthroplasty, shoulder resurfacing arthroplasty, revision shoulder arthroplasty

Exclusion Criteria:

* Inability to complete follow-up questionnaires
* Declining operative management
* No desire to return to golf postoperatively
* Medical problem that affects the patient's ability to play golf (e.g., angina, shortness of breath, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing joint replacement surgery who are self-reported golfers and have a desire to return to golf postoperatively
Sampling Method: Non-Probability Sample
Enrollment: 432 (Estimated)
Dates: Start 2023-01-09 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of return to golf following joint arthroplasty | Up to 1 year postoperatively
  Patients will be asked if they have returned to golf (putting, chipping, 9 holes, 18 holes, etc) following joint arthroplasty.

SECONDARY OUTCOMES:
Golf awareness after arthroplasty score | Up to 1 year postoperatively
  This questionnaire assesses awareness of the joint replacement while playing golf and engaging in specific golf activities. A higher score represents more awareness, whereas a lower score represents less awareness.
Hip Disability and Osteoarthritis Outcome Score for Joint Replacement (HOOS JR) | Up to 1 year postoperatively
  The HOOS JR measures overall hip health on a scale of 0-100, where 0 represents total hip disability and 100 represents perfect hip health. This will be administered specifically to patients undergoing hip arthroplasty.
Knee Injury and Osteoarthritis Outcome Score for Joint Replacement (KOOS JR) | Up to 1 year postoperatively
  The KOOS JR measures overall knee health on a scale of 0-100, where 0 represents total knee disability and 100 represents perfect knee health. This will be administered specifically to patients who undergo knee arthroplasty.
American Shoulder and Elbow Surgeons Shoulder Score (ASES) | Up to 1 year postoperatively
  The ASES measures shoulder function on a scale of 0-100, where 0 represents worse function and 100 represents best function. This will be administered specifically to patients who undergo shoulder arthroplasty.

CONTACTS AND LOCATIONS:
Locations (2):
- Hospital for Special Surgery, New York, New York, United States
- Royal Infirmary of Edinburgh, Edinburgh, United Kingdom